CLINICAL TRIAL: NCT03049072
Title: A Prospective Registry Study to Record Clinical Results and Side Effects of Ion Beam Therapy at MedAustron
Brief Title: Ion Therapy Patient Registry
Acronym: REGI-MA-002015
Status: Recruiting | Type: Observational
Sponsor: EBG MedAustron GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: REGI-MA-002015
Record Dates: First submitted 2017-01-13; First posted 2017-02-09 (Estimated); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Ion Beam Radiation Therapy for Tumor Patients
MeSH Terms: interventions — Protons

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years

GROUPS / COHORTS (1):
- Ion beam therapy: All patients treated with ion beam therapy at MedAustron who consent to the participation in the registry.
  Interventions: Radiation: Protons and Carbon Ions

INTERVENTIONS:
Radiation: Protons and Carbon Ions

SUMMARY:
The purpose of the study is the prospective and standardized data collection of patients treated with ion therapy at MedAustron.

DETAILED DESCRIPTION:
During and up to 10 years after radiation therapy data regarding tumor control and treatment response as well as acute and late toxicities will be collected at regular time intervals. Additionally quality of life and sociodemographic status will be assessed in all study patients and neurocognitive assessment will be performed in patients undergoing ion radiation of the brain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tumor disease treated with ion beam therapy at MedAustron
* Signed informed consent form

Exclusion Criteria:

* Comorbidities endangering treatment delivery or study compliance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with ion beam therapy at MedAustron
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
Therapy response | 10 years
  Therapy Response according to RECIST Version 1.1
Overall survival | 10 years
Progression-free survival | 10 years
Local progression-free survival | 10 years
Cause-specific survival | 10 years
Toxicity according to NCI CTCAE | 10 years
  Acute/late toxicity according to CTCAEv4.03, June 14,2010

SECONDARY OUTCOMES:
EORTC-QLQ-C30 | Through study completion, at 3, 5, and 10 years
  Patient-reported quality of life
EORTC-QLQ-BN20 | Through study completion, at 3, 5, and 10 years
  Patient-reported quality of life for brain cancer patients
EORTC-QLQ-PR25 | Through study completion, at 3, 5, and 10 years
  Patient-reported quality of life for prostate cancer patients
Neurocognitive test battery | Through study completion, at 3, 5, and 10 years
  Change in cognition from baseline to endpoint as measured by standardized subtests of test battery

CONTACTS AND LOCATIONS:
Overall Officials: Carola Lütgendorf-Caucig, MD MPH MBA, Principal Investigator — EBG MedAustron GmbH; Piero Fossati, MD MSc, Principal Investigator — EBG MedAustron GmbH
Locations (1):
- EBG MedAustron GmbH, Wiener Neustadt, Lower Austria, Austria